CLINICAL TRIAL: NCT06899516
Title: Project MILANO: Connections Between Patients With Brain Tumors and Their Pets: an Analysis of Concerns and Needs
Acronym: MILANO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN252025/CHUSTE
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Brain (Nervous System) Cancers
Keywords: Brain tumors; Glioma patients; Pet care; Emotional burden
MeSH Terms: conditions — Neurologic Manifestations; Neoplasms; Brain Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pet-owning brain tumour patients: To assess the concerns and needs of patients with brain tumors regarding their pets, in order to plan for the pets' future when their owners are hospitalized, unable to care for them due to their condition, or in the event of their death.
  Interventions: Other: The Lexington Attachment to Pets Scale (LAPS; Johnson, Garrity, & Stallones, 1992)

INTERVENTIONS:
Other: The Lexington Attachment to Pets Scale (LAPS; Johnson, Garrity, & Stallones, 1992) — The LAPS is a established tool for measuring the emotional bond between humans and their animal companions. Animal attachment is assessed according to three factors: the bond between owners and their dogs or cats, the closeness of the human-animal relationship, and the importance of the animal in the owner's life (Johnson et al., 1992). Higher scores indicate greater attachment.

SUMMARY:
Context and problem

In France, 61% of households own a pet, highlighting the significant role pets play in the daily lives. Patients diagnosed with brain tumors face specific challenges that may affect their ability to care their pets, including:

* Progressive neurological deficits (cognitive and/or motor), limiting their autonomy,
* A life-threatening prognosis.

In this context, the well-being of pets when their owner's health deteriorates becomes a critical concern. Indeed:

* Social isolation and the progressive loss of physical and cognitive abilities complicate pet care, particularly during prolonged hospitalizations or in the event of death,
* The lack of appropriate facilities and care solutions causes stress for pets, who are often unprepared for such transitions, and adds to the emotional burden on patients.

Why focus on patients with brain tumors?

* These patients have specific needs due to the rapid progression of their condition,
* A local study showed that 12% of patients with gliomas live alone, a significantly higher rate than in other cancer types. Patients who live alone are particularly exposed to issues related to their pet's future,
* Given the high morbidity and mortality associated with brain tumors, proactive planning for pet care is particularly urgent.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with a brain tumor.
* Patients who own at least one pet.

Exclusion Criteria:

* Patients who decline to participate in the study.
* Patients unable to complete the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a brain tumor who have one or more pets will be included.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
LAPS scale | Day 1
  The Lexington Pet Attachment Scale (LAPS) measures the percentage of patients who are concerned about their pets. Values range from zero to one hundred, with higher scores indicating greater concern for pets.

SECONDARY OUTCOMES:
Questionnaire | Day 1
  A questionnaire that measures the percentage of patients who need more information and details of resources and support systems to help them with their pets.

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ramirez, Md, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No